CLINICAL TRIAL: NCT04952714
Title: Renal Replacement Therapy With a Cytokine Absorption Filter (oXiris ®) in Patients With Septic Shock: a Case-control Study Nested in a Cohort
Brief Title: RRT With a Cytokine Absorption Filter (oXiris ®) in Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Clinica CES (Network)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Acta240Proy010
Record Dates: First submitted 2021-04-11; First posted 2021-07-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury; Septic Shock
Keywords: Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dynamic Cohort: Initially, participants who meet the inclusion criteria will be recruited to assemble a cohort of patients with sepsis and those who develop sepsis-induced acute kidney injury will be observed.
  Through a previously established and standardized management protocol, the treating team will prescribe renal replacement therapy by hemodiafiltration (CVVHDF) in the PrismaFlex device (Baxter), at a dose of 25 mL / Kg of PrismaSate dialysis solution (Baxter) and the removal filter oXiris® cytokines (Baxter) vs. the standard filter, for patients who require it, in the presence of a confirmed diagnosis of acute renal failure.
  Hemodynamic and ventilatory parameters will be monitored every 24 hours, and inflammatory parameters every 48 hours. A follow-up will be done at 28 days to establish mortality.
  Interventions: Device: Oxiris

INTERVENTIONS:
Device: Oxiris — Through a previously established and standardized management protocol, the treating team will prescribe renal replacement therapy by hemodiafiltration (CVVHDF) in the PrismaFlex device, at a dose of 25 mL / Kg of PrismaSate dialysis solutio and the removal filter oXiris® cytokines (Baxter) vs. the standard filter.

SUMMARY:
Acute kidney injury (AKI) is a common complication in critically ill patients. Multiple studies have reported evidence that the main cause of ARF is sepsis, as part of the Multiple Organ Dysfunction Syndrome: up to 50% of septic patients develop acute renal failure.

RRT continues to be the standard management for severe acute renal failure, especially in its continuous modality and applied to the septic patient, generally with hemodynamic instability.

The presence of SA-AKI (sepsis-associated acute kidney injury) is associated with short-term and long-term adverse events, which include: prolonged hospital stay, the development of chronic kidney disease (CKD), increased cardiovascular risk and increased risk of death. Its presence is even considered a factor with an independent association with mortality and has a higher fatality rate than ARF developed by another etiology.

Different clinical studies have been developed based on the addition of hemoadsorption membranes to RRT that, although they have not shown significant differences in the reduction of mortality, have impacted secondary outcomes such as the reduction of pro-inflammatory cytokines, decrease in vasopressor support requirements, decrease in serum lactate, significant improvement in the SOFA score, improvement in oxygenation indices and decrease in hospital stay. These benefits are presented without reports of adverse events associated with its use.

The oXiris® filter was recently developed: a single high permeability membrane capable of removing cytokines and endotoxins during renal support with the addition of antithrombotic properties. The experience of its use is limited to in vitro studies, case reports, retrospective cohorts and an RCT that provide consistent evidence of its benefits.

A longitudinal, bi-directional, observational analytical study is proposed. A case-control study nested in a dynamic cohort will be developed to determine the effect of the use of hemofiltration with a cytokine removal filter (oXiris®) on the decrease in mortality at 28 days of patients with acute kidney injury induced by sepsis. (SA-AKI), as well as the dose of vasopressor support, oxygenation parameters and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who enter the Intensive Care Unit of the CES Clinic during the recruitment period with:
* Diagnosis of septic shock of any origin according to the definition of the Sepsis-3 consensus.
* Acute renal injury according to the KDIGO 2012 classification that requires continuous renal replacement therapy and that its origin is presumed to be septic origin.
* In invasive ventilatory support.
* Informed consent previously filled out by a guardian.

Exclusion Criteria:

* Patients under 18 years of age and women in pregnancy or postpartum will be excluded.
* Chronic kidney disease that requires RRT on an outpatient basis before admission to the ICU.
* Contraindication to the use of heparins or another anticoagulant
* Dissent to escalate therapeutic measures
* Terminal or irrecoverable condition according to the criteria of the specialist in critical medicine and intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the institutional Intensive Care Unit (CES Clinic) with acute kidney injury induced by sepsis and requiring renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Effect of the use of hemofiltration with a cytokine removal filter (oXiris®) in the reduction in mortality at 28 days of patients with acute kidney injury induced by sepsis (SA-AKI).
Cardiovascular support | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Effect of using hemofiltration with a cytokine removal filter (oXiris®) in reducing the dose of vasopressor support (mcg/g/min) in patients with acute kidney injury induced by sepsis (SA-AKI).
Pulmonary support | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Effect of using hemofiltration with a cytokine removal filter (oXiris®) in improving the oxygenation parameters (PaO2/FiO2) in patients with acute kidney injury induced by sepsis (SA-AKI).
Inflammatory markers | Every 48 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Effect of using hemofiltration with a cytokine removal filter (oXiris®) in reducing inflammatory markers (CRP, Procalcitonin, IL-6) in patients with sepsis-induced acute kidney injury (SA-AKI).

SECONDARY OUTCOMES:
Demographic characteristics of patients with sepsis-induced acute kidney injury (SA-AKI) on renal replacement therapy treated in the Intensive Care Unit of the CES Clinic. | 28 days
  Demographic variables such as age (years), gender, body mass index (Kg / Mt2) and previous comorbid pathologies will be taken from the electronic medical record.
Cardiovascular status: Lactate | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Changes from baseline Lactate (mmol/L) measurements with the cytokine removal filter (oXiris®) vs. the standard filter.
Cardiovascular status: pH | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Changes from baseline pH measurements with the cytokine removal filter (oXiris®) vs. the standard filter.
Inflammatory status: IL-6 | Every 48 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Changes from baseline IL-6 (pg/mL) measurements with the cytokine removal filter (oXiris®) vs. the standard filter.
Inflammatory status: Procalcitonin | Every 48 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Changes from baseline Procalcitonin (ng/mL) measurements with the cytokine removal filter (oXiris®) vs. the standard filter.
Inflammatory status: CRP | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  Changes from baseline C-Reactive Protein (mg/dL) measurements with the cytokine removal filter (oXiris®) vs. the standard filter.
Describe the treatment characteristics of patients with sepsis-induced acute kidney injury (SA-AKI) on renal replacement therapy treated in the Intensive Care Unit of the CES Clinic. | Every 24 hours, from date of admission to the Intensive Care Unit until discharge from the ICU or death from any cause, whichever came first. Assessed up to 2 weeks.
  The parameters used in renal replacement therapy (anticoagulation, duration and time to start in days) will be taken from the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: David Yepes-Gómez, MD, MSc, Principal Investigator — Clinica CES
Locations (1):
- Clinica CES, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No